CLINICAL TRIAL: NCT01898832
Title: to Investigate the Maternal Serum IL-17 Levels in Pregnant Women With Intrahepatic Cholestasis of Pregnancy
Brief Title: Il-17 Levels in Intrahepatic Cholestasis of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Ayse Kirbas, ayse kirbas, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: zekai tahir burak- cholestasis
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2013-07

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: Cholestasis, pregnant, interleukin 17
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Cholestasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: None Retained — maternal venous ad umbilical cordon blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate maternal and fetal serum IL-17 levels in pregnant women with intrahepatic cholestasis of pregnancy and to find out if Th-17 cells have a role in progress of intrahepatic cholestasis of pregnancy.

DETAILED DESCRIPTION:
Intrahepatic cholestasis of pregnancy (ICP) is the most prevalent pregnancy-specific liver disease. It occurs mainly in the second or third trimester of pregnancy. It typically resolves after delivery spontaneously but it is associated with an increased risk of adverse fetal outcomes.

The cause of ICP is heterogeneous, pathophysiology is poorly understood and therapies have been empiric. Genetic predispositions, environmental influences, dietary factors and hormonal influences have been studied and cited in the literature.

Comparing with placebo, ursodeoxycholic acid (UDCA) has been shown improvement in treatment of pruritus in previous studies. S-adenosylmethionine, guar gum, activated charcoal, dexamethasone, cholestyramine, etc. are not effective in the treatment of symptoms.

CD4+ T cells are an essential regulators of immune responses and inflammatory diseases. They are also called chief of orchestra cells of immune system. The balance between T helper-(Th)1, Th-2 and Th-17 cells and their cytokinergic interaction are crucial for the response of the organism. Th17 and its specific cytokine IL-17 are responsible for pathogenesis of autoimmune diseases as autoimmune uveitis, experimental autoimmune encephalomyelitis in animal models and potentially also in human autoimmune diseases such as multiple sclerosis, Crohn's disease, rheumatoid arthritis, psoriasis, primary biliary cirrhosis. Recently, IL-17 targeted therapies (secukinumab, ixekizumab and brodalumab) are being studied in Phase III clinical trials to evaluate their overall efficacy and safety for certain autoimmune diseases.

Th-17 levels have been investigated in normal and abnormal pregnancies and results were incompatible with each other. Some researchers have said that the level of IL-17 increased during pregnancy but the others not.

Low serum IL-17 is associated with premature birth. Up-regulation of the IL-17 is associated with preeclampsia.

K. Harada et all. (2009) demonstrated that IL-17-positive cells are associated with the chronic inflammation of bile ducts in primary biliary cirrhosis(PBC). Also, some authors demonstrated that Th-17-related cytokines were increased significantly in patients with PBC.

Maho Ichikawa et all. presented a case of male newborn infant who showed progressive severe cholestasis with selectively high Levels of Serum IL- 17.

Based on all this information, we decided to investigate maternal and fetal serum IL-17 levels of pregnants with ICP and the effects of UDCA therapy on it and find out if Th-17 cells have a role in progress of ICP.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of ICP

-

Exclusion Criteria:

multiple pregnancies known chronic illness

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The pregnant women with intrahepatic cholestasis who admitted our clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
il-17 levels | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: ayse kirbas, md, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak, Ankara, Ankara, Turkey (Türkiye)